CLINICAL TRIAL: NCT02698306
Title: Comparison of the Use of Dexamethasone and Diclofenac Sodium in Immediate Post-Operative Care in Third Molar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Geral de Vila Penteado (Other Government)
Responsible Party: Principal Investigator, Fábio Ricardo Loureiro Sato, Principal Investigator, Hospital Geral de Vila Penteado
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HospitalGVP
Record Dates: First submitted 2016-02-09; First posted 2016-03-03 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Dexamethasone: Dexametasone 4mg tablet every 8/8hs for 3 days
  Interventions: Drug: Dexamethasone
- Diclofenac Sodium (Active Comparator): Diclofenac Sodium: Diclofenac Sodium 50 mg tablet every 8/8 hs for 3 days
  Interventions: Drug: Diclofenac Sodium

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone
  Other Names: Decadron
  Arms: Dexamethasone
Drug: Diclofenac Sodium — Diclofenac Sodium
  Other Names: Voltarem
  Arms: Diclofenac Sodium

SUMMARY:
The investigators will select 30 patients with symmetrical impaction of third molars, according to Pell and Gregory dental impaction classification, who would be submitted to two surgical procedures, right and left, and in both surgeries dexamethasone 8 mg was administered in the pre-surgery phase, and the use of dexamethasone (12 mg/day) for 3 days on one side and diclofenac sodium (150 mg/day) for 3 days on the other side was continued, in a randomized, double-blind and cross-over trial so that all patients acted as control of themselves (split-mouth). Other drugs used in postoperative period, rescue analgesic and antibiotic therapy will be identical for all patients. The analyzed variables will be the visual analogue pain scale (VAS), total number of consumed analgesics, swelling and trismus (objectively), which were statistically analyzed by means of Student's t-test.

DETAILED DESCRIPTION:
STUDY DESIGN

Clinical double-blind, randomized, split-mouth trial. This study was submitted to and approved by the Human Research Ethics Committees of Hospital Geral de Vila Penteado under CAA Protocol: 34824714.8.0000.5446.

MASKING AND RANDOMIZATION

To ensure that the patient, the main researcher, the surgeon and the statistician were unaware of what drug would be used postoperatively, dexamethasone (4 mg) and diclofenac sodium (50 mg) were prepared in capsules of the same color and size, stored in similar vials and coded as drug No. 1 or drug No. 2. The drugs used in different procedures were disclosed only after acquisition and analysis of all data. The randomization procedure will be performed by a researcher not involved in the evaluation of patients and surgeries, using sequentially numbered sealed envelopes. Each envelope had the combination of drugs to be used in the postoperative period, protocol 1 (with 1 drug) or protocol 2 (drug 2) and the side of surgery (right or left). For each enrolled patient, the researcher not involved in patient assessment and surgery opened the envelope, will inform the main researcher of the protocol to be used postoperatively, and the surgeon of the side to be operated. The second surgical procedure was performed on the contralateral side, using another medical protocol postoperatively, with an interval of two months between procedures. Thus, the patient, the surgeon and the main researcher did not know which medical protocol would be used postoperatively.

The methodology of this study sought to follow the rules of the new CONSORT 2010 Statement.

SURGICAL PROCEDURES AND DRUGS

Five minutes before surgery, patients will receive pre-operative drugs (Cefazoline1g/Dexamethasone 8 mg/100 ml of 0.9% saline solution) intravenously.

With the patient in the supine position on the operating table, the surgeon perform the extra and intra oral antisepsis with chlorhexidine 0.2% and anesthesia of the inferior alveolar, lingual, buccal, posterior superior alveolar and greater palatine nerves respecting the protocol described by Malamed, with lidocaine 2% and epinephrine 1:100,000, with a maximum volume of 9 ml. Initially, an incision was made at the alveolar crest along the mesial or distal aspect in the mandibular branch to reach the distolingual region of the second molar, followed by intrasulcular incision surrounding the second molar to the interdental area between the second and first molar. Afterwards, the surgeon will raise the mucoperiosteal flap, perform an osteotomy procedure (with a high speed engine, spherical surgical drills No. 8, conical drills 702, with copious irrigation with saline solution 0.9%), tooth sectioning of the crown and/or roots (with a high speed engine, zecrya surgical drill with copious irrigation and saline solution 0.9%) when indicated for the case, tooth dislocation, dental avulsion, curettage and filing and copious irrigation of the cavity with saline solution 0.9 %, absorbable polyglactin 910 suture (Vycril 4.0 - Ethicon Johnson & Johnson do Brasil Ltda. - São Paulo). Then, the surgeon will make an incision was made in the jaw tuberosity along the mesial to distal aspect in order to reach the distolingual region of the second molar, followed by intrasulcular incision surrounding the second molar to the interdental area between the second and first molar, raised the total mucoperiosteal flap, ostectomy (with chisel gouge), tooth luxation, dental avulsion, curettage and filing and copious irrigation of the cavity with saline solution 0.9%, absorbable polyglactin 910 wound suture. The duration of the surgery was noted in minutes from the time of completion of the first anesthesia to the time of final suture.

POST-OPERATIVE MANAGEMENT

After surgery, the researcher in charge will give instructions for local hemostatic measures, nutrition, wound cleaning, physical exertion restriction, dosage and gave the drugs to the patient according to research protocol.

Protocol 1: Amoxycillin (500mg) 8/8 hours for 7 days, drug 1 8/8 h for 3 days and as rescue drug, in case of pain, Dipyrone (500mg) that could be consumed within 4 / 4hours.

Protocol 2: Amoxycillin (500mg) 8/8 hours for 7 days, drug 2 8/8 h for 3 days and as rescue drug, in case of pain, Dipyrone (500mg) that could be consumed within 4 / 4hours.

CLINICAL ASSESSMENTS

For both sides, the elapsed time of the surgical procedure will be recorded, which started at the time of the anesthetic puncture and complete at the end of the last suture.

The pain will be measured from an analog scale from 0 to 10 corresponding to: 0 = no pain, 1 and 2 = MILD, (easily tolerated), 3 to 5 = MODERATE (tolerable discomfort), 6 to 8 = strong (discomfort difficult to tolerate) and 9 to 10 = VERY STRONG (unbearable), besides the pain score annotations at pre-set times (immediate postoperative period, 4 and 8 hours postoperatively).

The patient filled a control file where the total number of tablets consumed within 72 hours was recorded.

The swelling will be assessed by comparing the values of three facial lines: (1) the distance from the lateral corner of the eye to the gonial angle of the operated side; (2) the distance from the bottom edge of the tragus to the commissure of the mouth on the operated side; (3) the distance between the lower edge of the tragus to the soft pogonion of the operated side (Figure 1). In three different times, evaluating the preoperative values (time 1) with postoperative values 2nd day (time 2) and 7th day (time 3) after surgery, measured by the third researcher.

Trismus will be assessed by comparing the values of the distance between the incisal edges of the upper and lower central incisors measured by a millimeter ruler. In three different times, evaluating the preoperative values (time 1) with postoperative values 2nd day (time 2) and 7th day (time 3) after surgery.

ELIGIBILITY:
Inclusion Criteria:

- Patients had to have four third molars indicating the need for extraction and in any position of impact, as long as there was symmetry between the two sides.

Exclusion Criteria:

* Patients with a history of alcoholism, drug use, antihistamine drugs, antidepressants, cimetidine or any drug that could interfere with the painful sensitivity of the patient.
* Patients with systemic disorders such as diabetes, hypertension, heart disease, allergy to any component of the formula, sulfa drugs and also pregnant women, nursing mothers, persons experiencing dental fear and children were excluded.
* Patients who had pericoronitis and/or radiolucent images associated with the teeth to be extracted

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-03 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Pain assessed with a Visual Analog Scale | 1 week
Swelling measured by an scale in mm | 1 week
Mouth Opening measured by an scale in mm | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Fábio Ricardo L. Sato, PhD, Principal Investigator — Hospital Geral de Vila Penteado
Locations (1):
- Hospital Geral de Vila Penteado, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No